CLINICAL TRIAL: NCT04829591
Title: The Jordanian Heart Failure Registry (JoHFR)
Brief Title: A Multicenter Registry to Study the Characteristics and Outcomes of Jordanian Heart Failure Patients.
Acronym: JoHFR
Status: Completed | Type: Observational
Sponsor: Jordan Cardio Vascular Research Group (Other)
Responsible Party: Principal Investigator, Hadi Abu-Hantash, principle investigator and study chair, University of Jordan
Other Study IDs: JoCVRG
Record Dates: First submitted 2021-03-31; First posted 2021-04-02 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Heart Failure; Chronic Heart Failure; Acute Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: observational — Heart failure, non interventional

SUMMARY:
Heart Failure research registry is a collection of computerized information about individuals with heart failure. The database in this registry is obtained from several Jordanian medical centers which will represent an extremely valuable resource for epidemiological research on heart failure patients.

DETAILED DESCRIPTION:
Understanding the cause of Heart Failure (HF) and how the body will respond to it, is critical for an effective treatment. HF is a global problem with significant morbidity and mortality, despite improved understanding of the pathophysiology and a growing range of therapeutic options. Jordanian Heart Failure Registry (JoHFR) will be the first research project of heart failure prevalence in Jordan. It is undertaken by primary healthcare professionals with main aim to improve knowledge about the care of patients with HF. The investigators responsible for conducting this research are physicians and their teams who deal with heart failure patients in their outpatient and inpatient clinic centers including the public and private medical sectors in Jordan's medical community. Standards in the Hashemite kingdom of Jordan complies with the recognized good guideline directed medical practices internationally

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are 18 years or older with Heart Failure diagnosis as defined by internationally recognized guidelines.
2. Current residents of the Hashemite Kingdom of Jordan

Exclusion Criteria:

1. Patients who refuse or unable to sign a consent form.
2. Patient inability to follow up with provider

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients 18 years old and older with HF will be recruited from all over Jordan , resulting in an initial sample estimate of approximately 4000 patients.
Sampling Method: Non-Probability Sample
Enrollment: 2219 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Cardiovascular death | 12 months
  The main objective of the JoHFR is to obtain reliable estimate of rates of cardiovascular death and or hospitalization for decompensated heart failure

SECONDARY OUTCOMES:
worsening kidney function | 12 months
  as compared to baseline eGFR

CONTACTS AND LOCATIONS:
Overall Officials: Hadi M Abu-Hantash, MD,MSc, Study Chair — Interventional Cardiovascular Innovation group
Locations (1):
- Farah Medical Campus, Amman, Jordan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Joseph P, Dokainish H, McCready T, Budaj A, Roy A, Ertl G, Gomez-Mesa JE, Leong D, Ezekowitz J, Hage C, Lanas F, Maggioni AP, Sliwa K, Zhu J, Rouleau J, Balasubramanian K, Yusuf S; G-CHF Investigators. A multinational registry to study the characteristics and outcomes of heart failure patients: The global congestive heart failure (G-CHF) registry. Am Heart J. 2020 Sep;227:56-63. doi: 10.1016/j.ahj.2020.06.002. Epub 2020 Jun 6. PMID 32679282
- [Background] Savarese G, Vasko P, Jonsson A, Edner M, Dahlstrom U, Lund LH. The Swedish Heart Failure Registry: a living, ongoing quality assurance and research in heart failure. Ups J Med Sci. 2019 Jan;124(1):65-69. doi: 10.1080/03009734.2018.1490831. Epub 2018 Aug 9. PMID 30092697
- [Background] Crespo-Leiro MG, Anker SD, Maggioni AP, Coats AJ, Filippatos G, Ruschitzka F, Ferrari R, Piepoli MF, Delgado Jimenez JF, Metra M, Fonseca C, Hradec J, Amir O, Logeart D, Dahlstrom U, Merkely B, Drozdz J, Goncalvesova E, Hassanein M, Chioncel O, Lainscak M, Seferovic PM, Tousoulis D, Kavoliuniene A, Fruhwald F, Fazlibegovic E, Temizhan A, Gatzov P, Erglis A, Laroche C, Mebazaa A; Heart Failure Association (HFA) of the European Society of Cardiology (ESC). European Society of Cardiology Heart Failure Long-Term Registry (ESC-HF-LT): 1-year follow-up outcomes and differences across regions. Eur J Heart Fail. 2016 Jun;18(6):613-25. doi: 10.1002/ejhf.566. PMID 27324686
- [Background] Bergethon KE, Ju C, DeVore AD, Hardy NC, Fonarow GC, Yancy CW, Heidenreich PA, Bhatt DL, Peterson ED, Hernandez AF. Trends in 30-Day Readmission Rates for Patients Hospitalized With Heart Failure: Findings From the Get With The Guidelines-Heart Failure Registry. Circ Heart Fail. 2016 Jun;9(6):10.1161/CIRCHEARTFAILURE.115.002594 e002594. doi: 10.1161/CIRCHEARTFAILURE.115.002594. PMID 27301467

DOCUMENTS (2):
  • Study Protocol (2021-04-17): https://cdn.clinicaltrials.gov/large-docs/91/NCT04829591/Prot_000.pdf
  • Informed Consent Form (2021-04-17): https://cdn.clinicaltrials.gov/large-docs/91/NCT04829591/ICF_001.pdf